CLINICAL TRIAL: NCT07163442
Title: One-year Results of Bioidentical Hormone Replacement Therapy in Postmenopausal Women
Brief Title: Bioidentical Hormone Replacement Therapy in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, dr, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasatrehmENA
Record Dates: First submitted 2025-08-19; First posted 2025-09-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Hormon Replacement Terapy
Keywords: post-menopausal; hormone replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 107 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grup:1 group not taking postmenopausal hormones: postmenopausal women who have been in menopause for at least 1 year and have not taken any hormone supplements
- grup 2: Patients who have been receiving HRT for 1 year: Patients who have been using HRT for at least 1 year since the onset of menopause

SUMMARY:
The aim of this observational study is to investigate the effects of bioidentical HRT over a 1-year period in postmenopausal women receiving transdermal estradiol and, when necessary, progesterone. The main question the study aims to answer is:

Does bioidentical hormone replacement therapy, when used long-term in postmenopausal women, reduce the negative effects of menopause compared to women who do not receive it? Participants who were already receiving bioidentical transdermal estradiol and micro-dose progesterone as part of their regular medical care under postmenopausal hormone therapy were compared to a group not receiving such therapy over a one-year period, with measurements taken of bone densitometry, mammography, blood lipid parameters (HDL, LDL, VLDL, total cholesterol), and HbA1c levels.

DETAILED DESCRIPTION:
The aim of this observational study is to investigate the effects of bioidentical HRT over a 1-year period in postmenopausal women receiving transdermal estradiol and, when necessary, progesterone. The main question the study aims to answer is:

Does bioidentical hormone replacement therapy, when used long-term in postmenopausal women, reduce the negative effects of menopause compared to women who do not receive it? Participants who were already receiving bioidentical transdermal estradiol and micro-dose progesterone as part of their regular medical care under postmenopausal hormone therapy were compared to a group not receiving such therapy over a 1-year period, with measurements taken of bone densitometry, mammography, blood lipid parameters (HDL, LDL, VLDL, total cholesterol), and HbA1c levels. Additionally, they were asked to complete a questionnaire aimed at assessing the severity of vasomotor symptoms during menopause. The patients were divided into two groups. Group 1 consisted of women who had been in menopause for one year and had never taken HRT, while Group 2 consisted of women who had been in menopause for one year or more and were using transdermal bioidentical HRT and micronized progesterone. The values of these two groups were compared to evaluate the effect of HRT

ELIGIBILITY:
Inclusion Criteria:

* Being in menopause for a year
* being on hormone replacement therapy

Exclusion Criteria:

* taking HRT in addition to the drugs monitored in the study
* having a hormone-secreting endocrine disorder
* having endocrine cancer(breast cancer...)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since our study evaluates postmenopausal processes, it can only be conducted on women.
Study Population: Patients who have been in menopause for at least 1 year and do not have endocrine or metabolic disorders that alter hormone levels.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
bone mineral densitometry | From enrollment to the end of treatment at one-year"
  In bone mineral densitometry, the T and Z scores of the left femur and spine will be examined. Values above -1.5 are considered normal, values between -1.5 and -2.5 indicate osteopenia, and values below -2.5 indicate osteoporosis.

SECONDARY OUTCOMES:
mammography report | From enrollment to the end of treatment at one-year"
  B-RADS scores will be obtained from patients' mammography reports. This score ranges from 0 to 5.
  Category 0: Additional imaging is needed. Category 1: Normal findings. Category 2: Definitely benign findings. Category 3: Probably benign findings. Category 4: Suspicious findings. Category 5: High probability of malignant findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.

REFERENCES:
- [Result] Kissinger D. Hormone replacement therapy perspectives. Front Glob Womens Health. 2024 May 20;5:1397123. doi: 10.3389/fgwh.2024.1397123. eCollection 2024. PMID 38832110